CLINICAL TRIAL: NCT02369601
Title: Clinical Evaluation of PRO-MComplete as an Aid in Determination of Rupture of Fetal Membranes
Brief Title: PROMComplete for Determination of Rupture of Fetal Membranes
Acronym: (PROMComplete
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pro-Lab Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: PROMC001
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Fetal Membranes, Premature Rupture
Keywords: amniorrhexis; Ruptured membranes; Alfa-fetoprotein
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: non- intervention study — Study design is non-interventional. Patient therapy will not be affected by study participation.

SUMMARY:
Premature rupture of membranes refers to the rupture of the fetal membranes prior to the onset of labor. Premature rupture of membranes is associated with a number of neonatal and maternal complications including an increased incidence of perinatal mortality and intra-amniotic infection. There is a need for improved diagnostic testing because of limitations of the current methods.

PRO-MComplete is an immunochromatographic test that detects insulin growth factor binding protein 1 and alpha-fetoprotein in vaginal fluid as an indicator of membrane rupture.

DETAILED DESCRIPTION:
Premature rupture of membranes (PROM) complicates approximately 8 % of pregnancies and is generally followed by the prompt onset of spontaneous labor and delivery. Preterm PROM complicates only 2 % of pregnancies but is associated with 40% of preterm deliveries and can result in significant neonatal morbidity and mortality (ACOG 2007). Intraamniotic infection has been shown to be commonly associated with preterm PROM, especially at earlier gestational ages (ACOG 2013). Currently, the diagnosis of PROM is based primarily on the patient's history and physical examination. The diagnosis of membrane rupture typically is confirmed by the visualization of amniotic fluid passing from the cervical canal and pooling in the vagina; a basic pH test of vaginal fluid; or arborization (ferning) of dried vaginal fluid, which is identified under microscopic evaluation (ACOG 2013).

The classic clinical presentation of PROM is a sudden "gush" of clear or pale yellow fluid from the vagina. However, many women describe intermittent or constant leaking of small amounts of fluid or just a sensation of wetness within the vagina or on the perineum (WHEC 2009).

However, the diagnosis of PROM is difficult if there is a slow fluid leak or any bleeding, or when the classic "gush of fluid "does not occur (Bornstein 2006).

Although ultrasonographically guided transabdominal instillation of indigo carmine dye and observation for fluid passage transvaginally is designated an "unequivocal" diagnostic method for confirmation of membrane rupture, this invasive test carries increased maternal and fetal risk (Mercer 2004). The absence of a non-invasive "gold standard" for the diagnosis of PROM has led to technically advanced biochemical markers for improved diagnosis (El-Messidi, 2010).

The AmniSure ROM (Rupture of Membranes) test received Food and Drug Administration 510(k) marketing clearance in 2003. A comparison study of AmniSure versus standard diagnostic methods for detection of ROM in 203 pregnant women suspected of ROM reported that the AmniSure test was highly accurate (sensitivity = 98.9 %, specificity = 100 %, and negative predictive value [NPV] = 99.1 %) in diagnosing ROM (Cousins et al, 2005). Test performance was calculated by comparing AmniSure results against clinical history, nitrazine and fern results, presence of pooling, ultrasound (US) evidence of oligohydramnios, and findings from repeated examinations.

Chen and Dudenhausen (2008) compared 2 rapid strip tests for the detection of amniotic fluid, based on the detection of insulin-like growth factor-binding protein-1 (IGFBP-1) and of PAMG-1. Samples of amniotic fluid were taken in 20 pregnant women between 31 3/7 and 41 2/7 gestational weeks at elective cesarean section before delivery of the newborn. These samples were diluted with 0.9 % saline solution in a dilution series down to concentrations of 1:320. Immunoassay strip tests were then compared in their ability to detect remaining concentrations of amniotic fluid. In 5 cases, both test methods showed the same results. In all remaining 15 cases, the test based on PAMG-1 proved to be superior by detecting amniotic fluid at least at one descending concentration below the test based on IGFBP-1.

PRO-MComplete proposes an alternative tool for adjuvant diagnosis of PROM by identification of Insulin-Like Growth Factor Binding Protein1 and Alpha Feto- Protein (AFP). The addition of AFP is projected to increase the sensitivity and specificity of PRO-MComplete over IGFBP-1 alone.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided verbal and written informed consent to participate in the study.
2. 20-42 weeks of gestation.
3. Subject presents with signs and/or symptoms of premature rupture of membranes.
4. Subject age 18 (years) or older

Exclusion Criteria:

1. Placenta Previa
2. Presenting with vaginal bleeding
3. Intravaginal ultrasound with presence of transducer gel
4. Active labor
5. Imminent delivery
6. Intercourse within 24 hours
7. Cord prolapse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will be women presenting with signs, symptoms or suspicion of membrane rupture at 20 to 42 weeks gestation.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
accuracy of Pro-mcomplete vs conventional testing for ruptured fetal membranes | up to 20 weeks
  All eligible subjects will be evaluated clinically and will be tested with appropriate reference tests as well as the PRO-MComplete test. Subjects tested with Pro-mcomplete will be followed until delivery of index pregnancy. Final subject evaluation will occur with index delivery.

SECONDARY OUTCOMES:
Occurrence of discordant examination | up to 20 weeks
  Documentation of frequency of device and clinical examination incongruent results. Pregnancy outcomes will be reviewed for all test subjects, not just the test incongruent cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rae, Study Director — Pro-Lab Diagnostic VP; Hector Chapa, M.D., Principal Investigator — Methodist Medical Center Dallas
Locations (6):
- United States (6):
  - University of Alabama Hospital, Birmingham, Alabama
  - Indiana University, Indianapolis, Indiana
  - Methodist Hospital Dallas, Dallas, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
  - Christus Santa Rosa Westover Hills, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah

REFERENCES:
- [Background] ACOG Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 80: premature rupture of membranes. Clinical management guidelines for obstetrician-gynecologists. Obstet Gynecol. 2007 Apr;109(4):1007-19. doi: 10.1097/01.AOG.0000263888.69178.1f. PMID 17400872
- [Background] Practice bulletins No. 139: premature rupture of membranes. Obstet Gynecol. 2013 Oct;122(4):918-930. doi: 10.1097/01.AOG.0000435415.21944.8f. PMID 24084566
- [Background] Women's Health and Education Center, Obstetrics: Premature Rupture of Membranes: Diagnosis and Management. http://www.womenshealthsection.com/content/obs/obs021.php3 Accessed July 13, 2009
- [Background] Bornstein J, Geva A, Solt I, Fait V, Schoenfeld A, Shoham HK, Sobel J. Nonintrusive diagnosis of premature ruptured amniotic membranes using a novel polymer. Am J Perinatol. 2006 Aug;23(6):351-4. doi: 10.1055/s-2006-947159. Epub 2006 Jul 13. PMID 16841279
- [Background] Mercer BM. Preterm premature rupture of the membranes: diagnosis and management. Clin Perinatol. 2004 Dec;31(4):765-82, vi. doi: 10.1016/j.clp.2004.06.004. PMID 15519427
- [Background] El-Messidi A, Cameron A. Diagnosis of premature rupture of membranes: inspiration from the past and insights for the future. J Obstet Gynaecol Can. 2010 Jun;32(6):561-569. doi: 10.1016/S1701-2163(16)34525-X. PMID 20569537
- [Background] Cousins LM, Smok DP, Lovett SM, Poeltler DM. AmniSure placental alpha microglobulin-1 rapid immunoassay versus standard diagnostic methods for detection of rupture of membranes. Am J Perinatol. 2005 Aug;22(6):317-20. doi: 10.1055/s-2005-870896. PMID 16118720
- [Background] Chen FC, Dudenhausen JW. Comparison of two rapid strip tests based on IGFBP-1 and PAMG-1 for the detection of amniotic fluid. Am J Perinatol. 2008 Apr;25(4):243-6. doi: 10.1055/s-2008-1066876. PMID 18548399